CLINICAL TRIAL: NCT04544449
Title: A Phase III Multicenter, Randomized, Double-Blind, Double-Dummy, Parallel-Group Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Ocrelizumab in Adult Patients With Primary Progressive Multiple Sclerosis.
Brief Title: A Study to Evaluate the Efficacy and Safety of Fenebrutinib Compared With Ocrelizumab in Adult Participants With Primary Progressive Multiple Sclerosis
Acronym: FENtrepid
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GN41791; 2019-003919-53 (EudraCT Number); 2022-502611-10-00 (EU CTIS Number)
Record Dates: First submitted 2020-09-04; First posted 2020-09-10 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive | interventions — fenebrutinib; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Sponsor will also be blinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fenebrutinib (Experimental): Participants will receive oral fenebrutinib and intravenous (IV) ocrelizumab-matching placebo.
  Interventions: Drug: Fenebrutinib; Drug: Placebo matched to ocrelizumab
- Ocrelizumab (Active Comparator): Participants will receive intravenous (IV) ocrelizumab and oral fenebrutinib-matching placebo.
  Interventions: Drug: Ocrelizumab; Drug: Placebo matched to fenebrutinib

INTERVENTIONS:
Drug: Fenebrutinib — Participants will receive fenebrutinib.
  Arms: Fenebrutinib
Drug: Ocrelizumab — Participants will receive ocrelizumab.
  Arms: Ocrelizumab
Drug: Placebo matched to ocrelizumab — Participants will receive ocrelizumab-matching placebo.
  Arms: Fenebrutinib
Drug: Placebo matched to fenebrutinib — Participants will receive fenebrutinib-matching placebo
  Arms: Ocrelizumab

SUMMARY:
A study to evaluate the efficacy and safety of fenebrutinib on disability progression in adult participants with Primary Progressive Multiple Sclerosis (PPMS). All eligible participants will be randomized 1:1 to either daily oral fenebrutinib (and placebo) or intravenous (IV) ocrelizumab (and placebo) in a blinded fashion through an interactive voice or web-based response system (IxRS). 985 participants were enrolled and recruited globally. Participants who discontinue study medication early or discontinue from the study will not be replaced. The Open-Label Extension (OLE) phase is contingent on a positive benefit-risk result in the Primary Analysis of the study.

ELIGIBILITY:
Inclusion Criteria:

* For sites in Germany and Italy only, enrollment is restricted to participants aged 46-65 years
* A diagnosis of PPMS in accordance to the revised 2017 McDonald Criteria (Thompson et al. 2018).
* Disability progression in the 12 months prior to screening.
* Expanded Disability Status Scale (EDSS) score from 3.0 to 6.5 inclusive at screening.
* Pyramidal functional subscore >=2 at screening.
* For participants currently receiving proton pump inhibitors (PPIs), H2-receptor antagonists (H2RAs), symptomatic treatment for MS (e.g. fampridine, cannabis) and/or physiotherapy: treatment at a stable dose during the screening period prior to the initiation of study treatment and plans to remain at a stable dose for the duration of study treatment.
* Neurologically stable for at least 30 days prior to randomization and baseline assessments.
* Ability to complete the 9-Hole Peg Test (9-HPT) for each hand in <240 seconds.
* Ability to perform Timed 25-Foot Walk Test (T25FWT) in <150 seconds.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

OLE Inclusion Criteria:

* Completed the Double-Blind Treatment (DBT) phase of the study (remaining on study treatment; no other Disease-Modifying Therapy (DMT) administered) and who, in the opinion of the investigator, may benefit from treatment with fenebrutinib.
* For female participants of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating eggs.
* For male participants: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and refrain from donating sperm.

Exclusion Criteria:

* For participants enrolled in Germany and in Italy only: Presence of gadolinium-enhancing lesions on T1-weighted MRI (T1Gd +) lesion on the screening MRI
* Any known or suspected active infection (excluding onychomycosis) at screening, including but not limited to a positive screening test for Hepatitis B and C, an active or latent or inadequately treated infection with tuberculosis (TB), a confirmed or suspected progressive multifocal leukoencephalopathy (PML).
* Participants with a previous history of a serious Infusion-Related Reaction (IRR) (Common Terminology Criteria for Adverse Events [CTCAE] Grade >= 4) and/or any hypersensitivity reaction to ocrelizumab.
* History of cancer including hematologic malignancy and solid tumors within 10 years of screening. Exceptions: Basal/squamous cell carcinoma of skin cured by excision. In situ carcinoma of the cervix successfully treated by curative therapy >1 year prior to screening.
* Known presence of other neurological disorders, that could interfere with the diagnosis of MS or assessments of efficacy or safety during the study, clinically significant cardiovascular, psychiatric, pulmonary, renal, hepatic, endocrine, metabolic or gastrointestinal disease.
* Presence of cirrhosis (Child-Pugh Class A, B, or C)
* Chronic liver disease unless considered stable for >6 months
* Acute liver disease
* Any concomitant disease that may require chronic treatment with systemic corticosteroids, immunosuppressants or specific medication that could impact the primary evaluation of the study.
* History of alcohol or other drug abuse within 12 months prior to screening.
* Female participants who are pregnant or breastfeeding or intending to become pregnant during the study or 6 or 12 months (as applicable from the local label for ocrelizumab) after final dose of study drug.
* Male participants intending to father a child during the study or for 28 days after final dose of study drug.
* Lack of peripheral venous access.
* Any previous treatment with immunomodulatory or immunosuppressive medication without an appropriate washout period.
* Receipt of a live or live-attenuated vaccine within 6 weeks prior to randomization.
* Immunocompromised state, history of primary or secondary (non-drug related) immunodeficiency, or history of transplantation or antirejection therapy
* Known bleeding diathesis, anemia, or history of hospitalization or transfusion for gastrointestinal (GI) bleed
* Any previous treatment with cladribine, mitoxantrone, daclizumab, alemtuzumab, or cyclophosphamide

OLE Exclusion Criteria:

* Chronic liver disease unless considered stable for > 6 months
* Acute liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 985 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2025-09-17 (Actual); Study Completion 2027-07-21 (Estimated)

PRIMARY OUTCOMES:
Time to Onset of Composite 12-week Confirmed Disability Progression (cCDP12) | Minimum of 120 weeks

SECONDARY OUTCOMES:
Time to Onset of Composite 24-week CDP (cCDP24) | Minimum of 120 weeks
Time to Onset of 12-week CDP (CDP12) | Minimum of 120 weeks
Time to Onset of 24-week CDP (CDP24) | Minimum of 120 weeks
Percentage Change in Total Brain Volume Assessed by Magnetic Resonance Imaging (MRI) | From Week 24 to Week 120
Change from Baseline in Participant-Reported Physical Impacts of Multiple Sclerosis (MS) Measured by the Multiple Sclerosis Impact Scale, 29-Item [MSIS-29] Physical Scale | Baseline, Weeks 12, 24, 36, 48, 60, 72, 84, 96, 108 and 120
  The MSIS-29, Version 2 is a 29-item patient-reported measure of the physical and psychological impacts of MS. Participants are asked to rate how much their functioning and well-being has been impacted over the past 14 days on a 4-point scale, from "Not at all" (1) to "Extremely" (4). The physical score is the sum of items 1-20, which is then transformed to a 0-100 scale. The psychological score is the sum of items 21-29, transformed to a 0-100 scale. Higher scores indicate a greater impact of MS.
Time to Onset of 12-week Confirmed 4-point Worsening in Symbol Digit Modality Test (SDMT) Score | Minimum of 120 weeks
  The SDMT is used for detecting the presence of cognitive impairment and changes in cognitive functioning over time and in response to treatment. The SDMT is brief, easy to administer test, and involves a simple substitution task. Using a reference key, the examinee has 90 seconds to pair specific numbers with given geometric figures. Responses will be collected only orally, and administration time is approximately 5 minutes. The number of correct responses in 90 seconds will be considered the SDMT score. A decrease by 4 points on the SDMT score from baseline represents a clinically meaningful change in cognitive processing. The SDMT score ranges from 0 to 110. The higher the results, the better processing speed/working memory.
Percentage of Participants with Adverse Events (AEs) | Up to 4.7 years
Plasma Concentrations of Fenebrutinib at Specified Timepoints | Up to 4.7 years
Percent Change from Screening in Blood Neurofilament Light Chain (NfL) Levels | Up to Week 120

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (189):
- United States (43):
  - Alabama Neurology Associates, Homewood, Alabama
  - Sutter East Bay Medical Foundation, Berkeley, California
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Palo Alto Medical Foundation Research Center, Sunnyvale, California
  - University of Colorado Denver, Aurora, Colorado
  - Yale University School Of Medicine, Fairfield, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Neurology Associates PA, Maitland, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School Of Medicine, Baltimore, Maryland
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - Wayne State University, Detroit, Michigan
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Washington University, St Louis, Missouri
  - Cleveland Clinic Lou Ruvo, Las Vegas, Nevada
  - Hackensack U Med Ctr, Hackensack, New Jersey
  - Barnabas Health Ambulatory Care Center, Livingston, New Jersey
  - Jersey Shore University Medical Centre, Neptune City, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - Dent Neurological Institute, Amherst, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Atrium Health Neurosciences Institute ? Charlotte, Charlotte, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - UC Health, LLC., Cincinnati, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - Providence Brain and Spine Institute, Portland, Oregon
  - Neurology Clinic PC, Cordova, Tennessee
  - Hope Neurology, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Uni of Texas Health Science Center At Houston, Houston, Texas
  - Texas Institute for Neurological Disorders, Sherman, Texas
  - Evergreen MS Center, Kirkland, Washington
  - Swedish Medical Center, Seattle, Washington
  - West Virginia University, Morgantown, West Virginia
  - Medical College of Wisconsin, Inc., Milwaukee, Wisconsin
- Argentina (5):
  - Centro de Especialidades Neurológicas y Rehabilitación - CENyR, Buenos Aires
  - Focus CECIC, Buenos Aires
  - Instituto Reumatológico Strusberg, Córdoba
  - Fundacion Rosarina de Neurorehabilitacion, Rosario
  - Centro de Investigaciones Médicas Tucuman, San Miguel
- Australia (7):
  - Brain and Mind Research Institute, Camperdown, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - John Hunter Hospital, New Lambton, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Box Hill Hospital, Box Hill, Victoria
  - Austin Hospital, Heidelberg, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (2):
  - Kepler Universitätsklinikum GmbH - Neuromed Campus, Linz
  - Medizinische Universität Wien, Vienna
- Brazil (7):
  - Santa Casa de Misericordia, Belo Horizonte, Minas Gerais
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Núcleo de Pesquisa do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - IMV Pesquisa Neurológica, Porto Alegre, Rio Grande do Sul
  - Clinica Neurologica, Joinville, Santa Catarina
  - Centro de Pesquisas Clinicas, São Paulo, São Paulo
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro
- Bulgaria (2):
  - UMHAT Dr. Georgi Stranski, Pleven
  - Multiprofile Hospital for Active Treatment of Neurology and Psychiatry Sv. Naum EAD, Sofia
- Canada (10):
  - University of Alberta Hospital, Edmonton, Alberta
  - Fraser Health Authority - Fraser Health Multiple Sclerosis, Burnaby, British Columbia
  - University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre Uni Campus, London, Ontario
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Clinique NeuroOutaouais, Gatineau, Quebec
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Chile (2):
  - CeCim Biocinetic, Santiago
  - Clinica Alemana, Vitacura
- Colombia (3):
  - Organizacion Sanitas Internacional, Bogotá
  - Fundacion Clinica Valle del Lili, Cali
  - Instituto Neurologico de Colombia INDEC, Medellín
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus N
  - Rigshospitalet, Glostrup Municipality
- France (6):
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hopital Pierre Wertheimer, Bron
  - CHRU de Montpellier, Hopital Gui de Chauliac, Montpellier
  - Hopital Guillaume Et Rene Laennec, Nantes
  - Hôpital Pasteur, Nice
  - Hopitaux Universitaires de Strasbourg, Strasbourg
- Germany (7):
  - Charite - Universitatsmedizin Berlin, Berlin
  - Studienzentrum Dr. Bischof GmbH, Böblingen
  - Universitätsklinikum "Carl Gustav Carus", Zentrum für Klinische Neurowissenschaften, Dresden
  - Universitätsklinikum Freiburg, Klinik für Neurologie und Neurophysiologie, Freiburg im Breisgau
  - Klinikum rechts der Isar der TU Muenchen, München
  - Universitaetsklinikum Tuebingen, Tübingen
  - Deutsche Klinik für Diagnostik, Wiesbaden
- Greece (3):
  - Hospital Eginition, Athens
  - 401 Military Hospital of Athens, Athens
  - AHEPA Univ. General Hospital of Thessaloniki, Thessaloniki
- Hungary (5):
  - Clinexpert Kft., Budapest
  - S-Medicon Egeszsegugyi Szolgaltato Kft., Budapest
  - Budapesti Jahn Ferenc Dél-pesti Kórház és Rendel?intézet, Budapest
  - Markhot Ferenc Oktatokorhaz és Rendelointezet, Eger
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
- Israel (3):
  - Rambam Medical Center, Haifa
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - AOU Seconda Università degli Studi, Napoli, Campania
  - A.O.U. di Parma, Parma, Emilia-Romagna
  - Policlinico Tor Vergata Dip. Neuroscienze-Clinica Neurologica-UOSD Sclerosi Multipla, Rome, Lazio
  - Irccs A.O.U.San Martino Ist, Genoa, Liguria
  - IRCCS Ospedale San Raffaele, Milan, Lombardy
  - Ospedale Civile di Montichiari, Montichiari, Lombardy
  - IRCCS Istituto Neurologico Neuromed, Pozzilli, Molise
  - A.R.N.A.S. Civico Di Cristina Benfratelli, Palermo, Sicily
- Mexico (5):
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - Hospital Juarez de Mexico, Mexico City, Mexico CITY (federal District)
  - Grupo Médico Camino S.C., México, Mexico CITY (federal District)
  - Clinical Research Institute, Tialnepantla, Mexico
- University Clinic of Neurology, Skopje, North Macedonia
- Peru (3):
  - Hospital IV Alberto Sabogal Sologuren, Bellavista
  - Clinica Internacional, Lima
  - Instituto Nacional de Ciencias Neurológicas - Hospital Mogrovejo, Lima
- Poland (10):
  - Neurocentrum Bydgoszcz sp. z o.o, Bydgoszcz
  - Care Clinic, Katowice
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Med Polonia, Późna
  - Centrum Medyczne "MEDYK", Rzeszów
  - Nmedis sp. z o.o., Rzeszów
  - Centrum Medyczne NeuroProtect, Warsaw
  - Wro Medica, Wroclaw
  - SPSK nr 1, Zabrze
- Portugal (5):
  - Hospital de Braga, Braga
  - Hospital Santo Antonio dos Capuchos, Lisbon
  - Hospital de Santa Maria, Lisbon
  - Hospital Geral de Santo Antonio, Porto
  - Hospital de Sao Joao, Porto
- San Juan MS Center, Guaynabo, Puerto Rico
- Russia (11):
  - Krasnoyarsk State Medical Academy, Krasnoyarsk, Krasnoyarsk Krai
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - Federal center of brain research and neurotechnologies, Moskva, Moscow Oblast
  - City Clinical Hospital #24, Moskva, Moscow Oblast
  - National Center of Social Significant Disease, Saint Petersburg, Sankt-Peterburg
  - City Hospital #40 of Resort Administrative District, Saint Petersburg, Sankt-Peterburg
  - Sverdlovsk Regional Clinical Hospital 1, Yekaterinburg, Sverdlovsk Oblast
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - Regional Multiple Sclerosis Centre b/o CC ECM Neftyanik, Tyumen, Tyumen Oblast
  - Center of Cardiology and Neurology, Kirov
  - State Novosibirsk Regional Clinical Hospital, Novosibirsk
- Spain (9):
  - Complejo Hospitalario Universitario A Coruña (CHUAC), A Coruña, LA Coruna
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida, Lerida
  - Hospital Quiron de Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Puerta del Mar, Cadiz
  - Hospital Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga ? Hospital General, Málaga
  - Hospital Universitario Virgen Macarena, Seville
- Switzerland (2):
  - Universitätsspital Basel, Basel
  - Inselspital Bern Medizin Neurologie, Bern
- Turkey (Türkiye) (10):
  - Hacettepe University Medical Faculty, Ankara
  - Baskent Universitesi Ankara Hastanesi, Çankaya
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi, Istanbul
  - Sancaktepe Training and Research Hospital, Istanbul
  - Selcuk University Medical Faculty, Istanbul
  - Kocaeli University Hospital, Kocaeli
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis Univ. Med. Fac., Samsun
  - Karadeniz Tecnical Uni. Med. Fac., Trabzon
  - Van Yuzuncu Yil University Hospital, Van
- Ukraine (13):
  - CNPE City Clinical Hospital #3 of Chernivtsi City Council, Chernivtsi, Chernihiv Governorate
  - MNE Lviv Territorial Medical Association Clinical Hospital for Palliative Care, Lviv, Chernihiv Governorate
  - Medical Centre of PE First Private Clinic, Zhytomyr, Crimean Regional Governmenta
  - Ams of Ukraine, Kharkiv, Kharkiv Governorate
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporizhzhia, Kharkiv Governorate
  - MEDBUD, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - Salutem Medical Center, Vinnytsia, KIEV Governorate
  - Separated structural unit ?University hospital? of Dnipro State Medical University, Dnipro, Tavria Okruha
  - Regional Clinical Hospital, Ivano-Frankivsk
  - Volyn Regional Clinical Hospital, Lutsk
  - Odesa Regional Clinical Hospital, Odesa
  - Medical Clinical Research Center of Medical Center LLC Health Clinic, Vinnytsia
- United Kingdom (4):
  - Queen Elizabeth University Hospital, Glasgow
  - Charing Cross Hospital, London
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Morriston Hospital, Swansea

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing